CLINICAL TRIAL: NCT01170676
Title: Promoting Asthma Wellness in Rural Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Henry Ford Health System (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Martha Tingen, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HL092412 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-07-27 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
Keywords: asthma; smoking; teens
MeSH Terms: conditions — Asthma; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Puff City GA (Experimental): Puff City is an NHLBI-funded (C. Joseph, PI; Henry Ford Health System, Detroit, MI), web-based intervention that targets three key asthma management issues in youth: 1) smoking reduction or cessation in those who are smokers, 2) improving adherence to asthma controller medication use, and 3) improving compliance of carrying a rescue inhaler at all times for use at the first sign of asthma symptoms. Puff City Ga. is a replication study in the rural southeastern United States that adds biological assessments in addition to self-report data.
  Interventions: Behavioral: Puff City GA
- General Asthma Education (Active Comparator): Students will be directed to generic public websites on asthma and smoking that contain helpful information on general asthma management.
  Interventions: Behavioral: General Asthma Education

INTERVENTIONS:
Behavioral: Puff City GA — Puff City GA focuses on three areas of health behavior: 1) adherence to controller medications; 2) immediate availability of rescue medication; 3)smoking cessation/reduction.
  Other Names: Behavioral Puff City Ga.
  Arms: Puff City GA
Behavioral: General Asthma Education — Students will be directed to generic public websites on asthma and smoking that contain helpful information on general asthma management.
  Arms: General Asthma Education

SUMMARY:
This is a research study that compares the effectiveness of a web-based program (known as Puff City) and another web-based program (of internet sites such as the American Lung Association, American Academy of Asthma, Allergy, and Immunology, etc) that targets five key asthma management issues among rural youth:

1. Improving adherence to asthma controller medication use;
2. Improving compliance of carrying a rescue inhaler at all times for use at the first sign of asthma symptoms;
3. Improving inhaler technique;
4. Smoking reduction or cessation in those who are smokers; and
5. Avoidance of second-hand smoke exposure.

DETAILED DESCRIPTION:
A randomized control trial across three southeastern rural high schools comparing a web-based tailored intervention (known as Puff City) to web-based traditional control education sites.

ELIGIBILITY:
Inclusion Criteria:

* AA ethnicity
* in 9th - 11th grade of selected rural schools
* have an asthma diagnosis and/or asthma-like symptoms by screening eligible on the Lung Health Survey
* have access to a telephone or mobile phone
* being the parent of a student meeting the above criteria with whom the student resides the majority of the time.

Exclusion Criteria:

* Not meeting the above criteria.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Actual)
Dates: Start 2009-08; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Days of asthma symptoms; personal cigarette smoking and cessation; and days of school missed because of asthma, measured by self report | baseline, end of treatment, 6 months, 12 months

SECONDARY OUTCOMES:
Change in exhaled nitric oxide and active and passive smoke exposure, measured by salivary cotinine. | baseline, end of treatment, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martha S Tingen, PhD, Principal Investigator — Augusta University; Dennis R Ownby, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Jordan DM, Bush JS, Ownby DR, Waller JL, Tingen MS. The impact of traditional literacy and education on health literacy in adolescents with asthma. J Asthma. 2019 Aug;56(8):882-890. doi: 10.1080/02770903.2018.1494191. Epub 2018 Sep 5. PMID 29984589